CLINICAL TRIAL: NCT03426722
Title: Phase III Study of L-carnitine vs Placebo for the Treatment of Muscle Cramps After Imatinib in Patients With Gastrointestinal Stromal Tumors (GISTs) (Single-center Study)
Brief Title: L-carnitine vs Placebo for the Treatment of Muscle Cramps After Imatinib in Gastrointestinal Stromal Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMC1801
Record Dates: First submitted 2018-01-29; First posted 2018-02-08 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Gastrointestinal Stromal Tumors (GISTs)
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-carnitine (Active Comparator): L-carnitine 500mg three times daily (per oral)
  Interventions: Drug: L-carnitine
- Placebo (Placebo Comparator): Placebo 500mg three times daily (per oral)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-carnitine — * L-carnitine VS Placebo is randomized (1:1)
  * L-carnitine 500mg TID(PO),
  * First evaluation will be performed at 8 weeks and then unblinding will be done. If symptoms continue after treatment, dose escalation in L-carnitine group by 1000mg TID (PO). If symptoms continue after treatment in Placebo group, L-carnitine 500mg TID(PO) will be given.
  Arms: L-carnitine
Drug: Placebo — Placebo 500mg TID(PO)
  Arms: Placebo

SUMMARY:
we aim to evaluate the efficacy of L-carnitine for the treatment of muscle cramps after imatinib in patients with GIST and apply in the future.

DETAILED DESCRIPTION:
One of the most common side effects of imatinib treatment, muscle cramps occur in about 30% of patients with gastrointestinal stromal tumor (GIST) receiving treatment with imatinib.

It affects the quality of life (QoL) of patients and could also be a factor that affects compliance with treatment. Some studies suggest that L-carnitine may improve muscle cramps associated with cirrhosis or hemodialysis. However, the efficacy of L-carnitine for muscle cramps occurring after imatinib treatment has yet to be reported. Thus, we aim to evaluate the efficacy of L-carnitine for the treatment of muscle cramps after imatinib in patients with GIST and apply in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed GIST patients who are taking imatinib
2. Age 18years or older
3. Patients experienced muscle cramps for more than 8 times (pain of NRS > 4) or 4 times (pain of NRS >7) within last 4 weeks
4. Life expectancy > 6 months
5. ECOG performance status of 0-3

Exclusion Criteria:

1. Patients with renal disease receiving hemodialysis
2. Liver Cirrhosis patients with Child-Pugh class B or C
3. Patients with history of hypersensitivity to drugs including L-carnitine or nutritional supplements
4. Patients with history of spinal cord injury, peripheral vascular disease, or > Grade 2 peripheral sensory neuropathy
5. Patients with clinically significant electrolyte imbalances such as hypocalcemia, hypokalemia, and hypomagnesaemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who have occurrence of muscle cramps ( numeric rating scale score > 4) | 4 weeks
  Proportion of patients who have occurrence of muscle cramps ( numeric rating scale score > 4) decreased by less than 50% in 4 weeks excluding the first 4 weeks of drug administration
  *numeric rating scale scores(range, 0-10) -> higher score is worse outcome

SECONDARY OUTCOMES:
Change in average numeric rating scale scores of muscle cramps | 4 weeks
  Change in average numeric rating scale scores(range, 0-10) of muscle cramps in 4 weeks excluding the first 4 weeks of drug administration
  *numeric rating scale scores(range, 0-10) -> higher score is worse outcome
Rate of patients who have duration of muscle cramps (numeric rating scale score > 4) | 4 weeks
  Rate of patients who have duration of muscle cramps (numeric rating scale score > 4)
  that was decreased by more than 50% in next 4 weeks excluding the first 4 weeks of drug administration
  *numeric rating scale scores(range, 0-10) -> higher score is worse outcome
questionnaire(Quality of Life) | 4 weeks
  Evaluation of the change in the Quality of Life in 4 weeks
plasma concentration level | 1 year
  Concentration evaluation of L-carnitine
recurrence rate | 1 year
  Recurrence is defined as 1) frequency of muscle cramps (NRS > 4) becomes more than 50% of baseline and 2) frequency of muscle cramps (NRS > 4) get twice worse than most improved time (when evaluated every 4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chae H, Ryu MH, Ma J, Beck M, Kang YK. Impact of L-carnitine on imatinib-related muscle cramps in patients with gastrointestinal stromal tumor. Invest New Drugs. 2020 Apr;38(2):493-499. doi: 10.1007/s10637-019-00860-x. Epub 2019 Oct 18. PMID 31628586